CLINICAL TRIAL: NCT07233109
Title: Energy Expenditure and Neuromuscular Function in Young Adult Women With a Naturally Thin Build (LeanErgy)
Acronym: LeanErgy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RIPH2_GADEA_LeanErgy; 2025-A01848-41 (Other: ID-RCB)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Constitutional Thinness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Woman with constitutional thinness (Experimental): Women aged between 18 and 35 Signed consent form Member of or entitled to social security Body Mass Index ≤ 17.5 kg/m2 Stable weight (no variation of more than 2kg over the last 12 months) No eating disorders No signs of malnutrition according to blood tests for cortisol* and FT3* No secondary amenorrhea
  Interventions: Diagnostic Test: Evaluation of the maximum oxidation point of lipids; Diagnostic Test: Evaluation of the energy cost of walking; Diagnostic Test: Neuro-muscular assessments
- Normal-weight women (Experimental): Women aged between 18 and 35 Signed consent form Member of or entitled to social security Body Mass Index between 20 kg/m² and 25 kg/m² Stable weight (No variation of more than 2 kg over the last 12 months) No eating disorders No secondary amenorrhea
  Interventions: Diagnostic Test: Evaluation of the maximum oxidation point of lipids; Diagnostic Test: Evaluation of the energy cost of walking; Diagnostic Test: Neuro-muscular assessments

INTERVENTIONS:
Diagnostic Test: Evaluation of the maximum oxidation point of lipids — The Lipoxmax measurement will take place in the morning, on an empty stomach. It will consist of a submaximal incremental exercise comprising five stages of six minutes each, with loads determined based on the power output obtained during the maximum oxygen consumption test and corresponding to 25%, 35%, 45%, 55%, and 65% of theoretical VO2 max. During the last minute of each stage, continuous measurement of VO2 and VCO2 will be used to calculate the average QR and then calculate the respective oxidation rates of carbohydrates and lipids, followed by the lipid oxidation rate at each stage. The oxidation rate curve is parabolic in shape, and modeling this curve will determine the lipoxmax point and the percentage of VO2max at which this lipoxmax point is obtained.
Diagnostic Test: Evaluation of the energy cost of walking — The energy cost of walking for participants will be assessed once for the NP group and twice and randomized for the MC group. All participants will have their energy cost assessed based on their body weight, and so will be in the MC group with a mechanical overload applied to simulate a BMI of 20 kg/m² (normal weight). This overload will be simulated with a weight corresponding to the weight required to achieve this BMI.
  Energy expenditure and energy substrates will be assessed during the walking exercise using portable indirect calorimetry (MetaMax, Inc.).This one is of the classic methods for measuring resting energy expenditure. For this exercise, participants will have to remain seated at rest for 10 minutes and then standing at rest for 5 minutes before performing an incremental submaximal walking exercise on a treadmill, consisting of 5 stages of 6 minutes each: i) 0.75 m.s-1; ii) 1 m.s-1; iii) 1.25 m.s-1; ii) 1.5 m.s-1; iv) 2.25 m.s-1. Each stage will be separated by 5 min.
Diagnostic Test: Neuro-muscular assessments — Neuromuscular function will be assessed using isokinetic dynamometry. Neuromuscular function of the lower limb (knee flexion/extension) Neuromuscular function of the upper limb (elbow flexion/extension)

SUMMARY:
People with a low BMI (<17.5) are most often considered to have anorexia nervosa (AN). However, recent literature suggests that there is a category of individuals with the same low BMI who do not meet the diagnostic criteria for anorexia nervosa but who have specific differences that make them a separate entity: constitutional thinness (CM). Constitutional thinness differs from anorexia nervosa in several ways. First, unlike AN, CM individuals do not have eating disorders and express a strong desire to gain weight. Another difference concerns the menstrual cycle: without oral contraception, AN individuals experience amenorrhea, while CM individuals have regular menstrual cycles. Biological signs of malnutrition are also present in anorexia nervosa, whereas this is not the case in constitutional thinness. Indeed, concentrations of IGF1, free T3, and leptin are significantly reduced in AN compared to healthy subjects, whereas there is no significant difference between healthy subjects and CT. Finally, in terms of body composition, there is a significant difference in particular in the percentage of fat mass between MC and AM subjects, with the MC group having a significantly lower percentage of fat mass than the control subjects but significantly higher than the AM subjects. The clinical management of MC patients could involve nutritional management of patients but also management in the form of an Adapted Physical Activity intervention program. However, this type of program using physical activity and a nutritional approach must be based on a characterization of the energy profile and physical abilities of MC patients, which remains to be studied. Germain et al. proposed measuring the physical activity level of MC patients using Actiheart (a combination of heart rate and accelerometer) and compared it with that of normal-weight (NW) individuals, finding no difference between the groups. However, this analysis remains a secondary analysis of their study, as the statistical power and choice of tool are certainly not appropriate for this question. Our team recently conducted the Nutrilean project, which for the first time questioned the aerobic and muscular capacities of women with CM compared to their NP counterparts. While our results show lower force production capacity in CM patients, suggesting neuromuscular adaptations to the chronic mechanical unloading caused by CM rather than an impairment of contractile abilities themselves, this remains to be explored more specifically. Indeed, these differences disappeared after normalization to body weight or muscle mass, suggesting a reduced gross force production capacity, but probably reflecting a normal physiological adaptation to low body and muscle mass. It now appears necessary to carry out more specific neuromuscular analyses in order to better understand the mechanisms, adaptations, and/or potential neuromuscular dysfunctions in this population. Similarly, while the results do not appear to show any impairment in the aerobic capacity of CM, they do highlight a potential impairment in their energy efficiency during locomotion, which may also reflect an adaptation to chronic exposure to lower mechanical loads.

In this context and following on from the work carried out to date by our team, the main objective of this study is i) to compare the lipid oxidation capacity and energy cost of walking between MC and NP participants; ii) to explore the adaptations of this energy cost in MC women in response to mechanical overload.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 17.5 kg/m2
* 20 kg/m2 ≤ BMI ≤ 25 kg/m2

Exclusion Criteria:

* For women with Constitutional thinness :

  * Women under guardianship or deprived of their liberty by judicial or administrative decision
  * Women who are pregnant, breastfeeding, or likely to become pregnant
  * Women who engage in intense physical activity (more than 3 sessions of physical activity per week)
  * Abnormal levels of IGF-1, estradiol, free T3, cortisol, and leptin
  * For the MC group specifically: cases of thinness due to a suspected organic cause. This includes Marfan syndrome, identifiable by: personal or family history of degenerative aortic disease (aneurysm, dissection), ligamentous hyperlaxity, arachnodactyly
  * History or presence of a systemic condition likely to interfere with the physiological and metabolic parameters measured (e.g., diabetes, endocrine or metabolic disease)
  * Any acute or chronic disease that may influence the results (e.g., infections, tumors, inflammatory diseases)
  * Medical or surgical history deemed by the investigator to be incompatible with this study (e.g., muscular, neurological, or joint disorders, or contraindications to the application of a magnetic field, etc.) Presence of diabetes, and any other condition limiting the application of either strategy under trial
  * Use of medications that may interfere with the study results
  * Cardiovascular conditions (history of cardiovascular and/or neurovascular disease, as well as the presence of cardiovascular and/or neurovascular risk factors other than obesity/overweight, such as: high blood pressure, high cholesterol, diabetes, heart rhythm disorder, known carotid atherosclerosis, thrombophilia)
  * Surgery within the previous 3 months
  * Women excluded from another study
  * Regular tobacco or alcohol consumption
  * Specific diets likely to impact metabolism, influence biological parameters (FT3, cortisol in particular) or skew results (deficiencies, low calorie intake). This includes vegan, mono, ketogenic, and low-calorie diets, intermittent fasting, or diets requiring specific supplementation that may interfere with the endocrine system.

For women Normal-Weighted Women

* Women under guardianship or deprived of their liberty by judicial or administrative decision
* Women who are pregnant, breastfeeding, or likely to become pregnant.
* Women who engage in intense physical activity (more than 3 sessions of physical activity per week)
* History or presence of a systemic condition likely to interfere with the physiological and metabolic parameters measured (e.g., diabetes, endocrine or metabolic disorders)
* Any acute or chronic disease that may influence the results (e.g., infections, tumors, inflammatory diseases)
* Medical or surgical history deemed by the investigator to be incompatible with this study (e.g., muscular, neurological, or joint disorders, or contraindications to the application of a magnetic field, etc.)
* Presence of diabetes or any other condition limiting the application of either strategy under investigation
* Taking medications that may interfere with the study results
* Cardiovascular conditions (history of cardiovascular and/or neurovascular disease, as well as the presence of cardiovascular and/or neurovascular risk factors other than obesity/overweight, such as: high blood pressure, high cholesterol, diabetes, heart rhythm disorder, known carotid atherosclerosis, thrombophilia)
* Surgery within the previous 3 months
* Women excluded from another study
* Regular tobacco or alcohol consumption
* Specific diets likely to impact metabolism, influence biological parameters, or skew results (deficiencies, low calorie intake). This includes vegan, mono, ketogenic, and low-calorie diets, intermittent fasting, or diets requiring specific supplementation that may interfere with the endocrine system.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 36 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Energy cost | 4 months
  Indirect calorimetry (measurement of gas exchange)

SECONDARY OUTCOMES:
Maximum lipid oxidation point | 4 months
  Indirect calorimetry (measurement of gas exchange)
Perception of effort | 4 months
  Borg Scale (0: zero effort -10 maximum effort)
Isometric and dynamic strength | 4 months
  Measurement on an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire AME2P, Université Clermont Auvergne, Aubière, France

IPD SHARING:
Plan to Share IPD: Undecided